CLINICAL TRIAL: NCT00682747
Title: Randomized Phase II Trial of Hyperbaric Oxygen for the Treatment of Radiation-induced Xerostomia
Brief Title: Hyperbaric Oxygen for the Treatment of a Dry Mouth Which Occurred After Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Thomas Kuhnt (Other)
Collaborators: Verband Deutscher Druckkammerzentren (Unknown)
Responsible Party: Sponsor-Investigator, Thomas Kuhnt, Dr. med., Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKSH-037
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Radiation-induced Xerostomia
Keywords: xerostomia; hyperbaric oxygenation; radiotherapy
MeSH Terms: conditions — Xerostomia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBO (Experimental): 40 treatments with hyperbaric oxygen once per day, five days per week, 2.4 ATA, 100 % oxygen (10-15 minutes compression with air, 90 min of oxygen breathing - two 10 minutes break for breathing air after each 30 minutes of oxygen, 10 minutes decompression with oxygen)
  Interventions: Drug: Hyperbaric oxygen
- non HBO (No Intervention)

INTERVENTIONS:
Drug: Hyperbaric oxygen — 40 treatments with hyperbaric oxygen once per day, five days per week, 2.4 ATA, 100 % oxygen (10-15 minutes compression with air, 90 min of oxygen breathing - two 10 minutes break for breathing air after each 30 minutes of oxygen, 10 minutes decompression with oxygen
  Arms: HBO

SUMMARY:
The purpose of this study is to determine whether hyperbaric oxygen is effective in the treatment of a dry mouth that occured after radiotherapy for head and neck tumours.

ELIGIBILITY:
Inclusion Criteria:

* complaints of xerostomia (visual analogue scale)
* at least 6 months after radiotherapy of the head and neck region including all salivary glands with at least 50 Gy
* objective hyposalivation / xerostomia (at rest < 0,25 ml saliva per minute, stimulated < 0,1 ml saliva per minute)
* patient must have given written informed consent

Exclusion Criteria:

* prior radiotherapy was an intensity modulated radiotherapy
* prior hyperbaric oxygen therapy after radiotherapy
* conditions which might be an additional risk for the treatment with hyperbaric oxygen such as spontaneous pneumothorax within the last two years, surgery of the eardrum or the middle ear, acute infection of the upper airways, not adequately treated epilepsy, concurrent radio- or chemotherapy, hereditary spherocytosis, psychosis, lung emphysema, asthma, severe COPD, prior surgery of the thorax, pace maker
* myocardial infarction within the last 6 months
* drug therapy which might induce xerostomia
* known intolerance or hypersensitivity to Wrigley's Freident®
* pregnancy or breast-feeding women (for women aged less than 60 years a pregnancy test is mandatory)
* women of childbearing potential with unclear contraception. The following contraceptive methods are recommended: combined oral contraceptives or progesterone-only pill, hormone-dispensing or copper intra-uterine system, hormone patches, long-acting injections, vaginal ring
* treatment with other investigational drugs or participation in another clinical trial within 30 days prior to enrollment
* refusal of cooperation or consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
change of overall salivation (millilitre per minute over 5 minutes measured at rest and after provocation) in percentages | baseline compared with measures on day 28, 56 and 146

SECONDARY OUTCOMES:
Number of Adverse Events in all patients as a Measure of Safety and Tolerability | baseline until 4 weeks after end of study treatment
Xerostomia scores assessed by investigator according to Eisbruch et.al. | baseline compared with measures on day 28, 56 and 146
Improvement of symptoms/discomfort due to xerestomia assessed by the patient on a visual analogue scale | baseline compared with measures on day 28, 56 and 146
quality of life measures (EORTC QLQ-H&N 35) | baseline compared with measures on day 28, 56 and 146

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kuhnt, MD, Principal Investigator — University Hospital Rostock, Clinic for Radiotherapy
Locations (2):
- Germany (2):
  - Martin Luther University Halle-Wittenberg, Clinic for Radiotherapy, Halle
  - Druckkammerzentrum Traunstein, Traunstein